CLINICAL TRIAL: NCT02597998
Title: Metabolism and Pharmacokinetics of [14C]-BI 409306 After Administration of 25 mg [14C]-BI 409306 as Oral Solution in Healthy Male Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]-BI 409306 After Administration as Oral Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1289.26; 2015-001877-42 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2015-11-05 (Estimated); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy

ARMS (1):
- 14C-BI 409306 - 25 mg (Experimental): 14C-BI 409306 oral solution
  Interventions: Drug: 14C-BI 409306

INTERVENTIONS:
Drug: 14C-BI 409306
  Other Names: 14C-BI 409306 oral solution

SUMMARY:
The aim of this study is to assess the mass balance recovery from excreta of carbon 14 labelled BI409306 ([14C] BI 409306) in healthy, CYP2C19 genotyped subjects and to provide plasma, urine and faecal samples for metabolite profiling and structural identification.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male genotyped as CY2C19 poor metabolizer (PM) or extensive metabolizer (EM) according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP - Blood Pressure, PR - Pulse Rate), 12-lead ECG (Electrogardiogramm), and clinical laboratory tests. PM is defined as carrier of two non-functional alleles *2 and *3 of the CYP2C19 gene (diplotypes *2/*2; *2/*3; *3/*3). EM is defined as carrier of two functional alleles of the CYP2C19 gene (absence of *2, *3, *17; diplotype *1/*1).
2. Age of 30 to 65 years (incl.).
3. BMI (Body Mass Index) of 18.5 to 29.9 kg/m2 (incl.).
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.
5. A history of regular bowel movements (averaging 1 or more bowel movements per day; subjects with regular bowel movements of >3 per day will be excluded).
6. Subjects who are sexually active must use, with their partner, 2 approved methods of highly effective contraception from the time of IMP administration until 90 days after the last dose of IMP.

Exclusion criteria:

1. Any finding in the medical examination (including BP - Blood Pressure, PR - Pulse Rate or ECG - Electrocardiogramm) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders. Any significant history of ocular or eye disease.
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was an open-label, single-arm, single-dose Phase I trial with healthy male subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 14C-BI 409306 - 25 mg: Healthy subjects received one single dose of oral solution containing 25 milligram (mg) of [14C]-BI 409306 containing a radioactive dose of approximately 2.00 Megabecquerel (MBq), reconstituted in 50 milliliter (mL) solvent (5 mg/mL tartaric acid solution)
Period: Overall Study
Arm/Group | 14C-BI 409306 - 25 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects in the randomised set (RS) (RS included all subjects who were assigned a study subject number, whether treated or not) who received the study drug.
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance Recovery of Total Radioactivity in Urine and Faeces: Amount Excreted Within the Time Interval From 0 to the Time of the Last Quantifiable Data Point as a Percentage of the Administered Dose (fe0-tz) for Urine and Faeces
Description: Mass balance recovery of total radioactivity in urine and faeces: Amount excreted within the time interval from 0 to the time of the last quantifiable data point as a percentage of the administered dose (fe0-tz) for urine and faeces. Urine collection intervals: -17:00-0:00 hours before drug administration and, 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192 and 192-216 hours after drug administration. Faeces collection intervals: -17:00-0:00, 0-24, 24-48, 48-72, 72-96, 96- 20, 120-144, 144-168, 168-192 and 192-216 hours after drug administration.
Time Frame: Urine and faeces sample collection: 17 hours before and up to 216 hours after drug administration. The details are mentioned in description section.
Population: The pharmacokinetic parameter analysis set (PKS) included all subjects in the treated set (TS) who provided at least one primary or secondary pharmacokinetic endpoint value, which was not flagged for exclusion.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of dose administered
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
Percentage (%) of dose administered
  Urine | 84.0 (4.42)
  Faeces | 10.4 (10.5)
  Urine and Faeces | 94.4 (4.45)

2. Secondary Outcome: Maximum Measured Concentration of BI 409306 in Plasma (Cmax)
Description: Maximum measured concentration of BI 409306 in plasma (Cmax).
Time Frame: PK plasma samples were taken at: 2:00 (hour: minute) before drug administration and 0:10, 0:20, 0:30, 0:45, 1, 1:30, 2, 2:30, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168 hours after drug administration.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) / Litre (L)
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
nanomole (nmol) / Litre (L) | 275 (24.3)

3. Secondary Outcome: Maximum Measured Concentration of 14C-BI 409306 Related Radioactivity in Plasma (Cmax)
Description: Maximum measured concentration of 14C-BI 409306 related radioactivity in plasma (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) / Litre (L)
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
nanomole (nmol) / Litre (L) | 1600 (15.6)

4. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) for BI 409306 in Plasma
Description: Area under the concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) for BI 409306 in plasma.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hour(h) / Litre (L)
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
nanomole (nmol) * hour(h) / Litre (L) | 357 (36.8)

5. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) for 14C-BI 409306 Related Radioactivity in Plasma
Description: Area under the concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) for 14C-BI 409306 related radioactivity in plasma.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hour(h) / Litre (L)
Arm/Group | 14C-BI 409306 - 25 mg
Number analyzed (Participants) | 6
nanomole (nmol) * hour(h) / Litre (L) | 3560 (9.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration, up to 21 days
Description: Treated Set: (TS) This subject set includes all subjects in the randomized set who received [at least] one dose of study drug. This was the full analysis set population in the sense of ICH-E9.
Arm/Group | 14C-BI 409306 - 25 mg
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 14C-BI 409306 - 25 mg (N=6)
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.